CLINICAL TRIAL: NCT05228756
Title: Fitness Intervention Trial in Adults With Sickle Cell Disease (SCD Fit): A Feasibility Study-Homebase Program
Brief Title: SCD Fit Homebase Program
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving institution
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Foluso Joy Ogunsile, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 300008284
Record Dates: First submitted 2021-12-09; First posted 2022-02-08 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Cardiovascular Diseases; Sickle Cell Disease; Exercise
MeSH Terms: conditions — Cardiovascular Diseases; Anemia, Sickle Cell; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resistance Band exercise for Sickle Cell Disease (Other): Participants will complete 16 exercise session at home wearing an accelerometer
  Interventions: Other: Accelerometer

INTERVENTIONS:
Other: Accelerometer — Participants will complete 16 exercise sessions at home wearing an accelerometer

SUMMARY:
The purpose of this project is to develop novel approaches to promote health and longevity while enhancing quality of life among persons with Sickle cell disease (SCD). Therefore, investigators are aiming to adapt an evidence-based exercise intervention for adults with SCD informed by culturally- relevant and biologic factors.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a major public health concern as it is the most common inherited blood disorder in the US, affecting predominantly African Americans.1 SCD causes intermittent painful vaso-occlusion events, which lead to multi-organ damage, significant morbidity and early mortality.2 As a result, individuals with SCD often report poor quality of life, high rates of work absenteeism, and increased healthcare utilization with estimated annual US healthcare costs of 786 million.3-5 Historically, individuals with SCD did not live beyond 18 years of age, but patients are now living into the fifth decade of life due to advancements in care.6 Cardiopulmonary disease (CVD) has replaced acute SCD-related complications as the leading cause of death for adults with SCD.7 Specifically, SCD increases the risk for pulmonary hypertension and congestive heart failure, which in turns causes mortality.8 Currently, there are knowledge gaps related to prevention of cardiopulmonary complications in SCD. There are no validated therapies or strategies to modify cardiopulmonary disease for persons with SCD (compared to other conditions) resulting in a disparity in care. Exercise is associated with improved quality of life, reduced morbidity, and decreased mortality in patients with advanced CVD, but regular exercise has yet to be studied in this context in SCD.9,10 For this reason, there is a critical need to evaluate the impact of exercise to address CVD risk and to promote longevity in SCD.

Previously, providers discouraged exercise for patients with advanced CVD.11 However, recent data suggest exercise is not associated with increased risk in this population.12 In non-SCD, advanced CVD, exercise training in cardiac rehabilitation is now considered an adjunctive tool to decrease chronic inflammation, improve CVD outcomes, and decrease mortality.10 Similarly, moderate-intensity exercise regimens can be completed in SCD without adverse complications.13 Mirroring the success of exercise therapy in CVD, there is potential for efficacy as a therapeutic tool in SCD to decrease inflammation, aid vascular endothelium remodeling, and improve endorgan dysfunction.14 Sterile inflammation secondary to chronic hemolysis is a well-characterized pathogenetic mechanism that occurs in the development of SCD cardiopulmonary disease.15 Regular exercise could modify CV disease progression in SCD by targeting inflammation that leads to microvascular damage.

In preparation for this project, we collected preliminary quantitative data in 69 adults with SCD; two-thirds of adults report physical inactivity, poor fitness, and exercise capacity - deficits that lead to poor CV outcomes and early mortality.16,17 We also found that adults with SCD have positive attitudes towards exercise and prefer individualized home-based programs but indicate an overall lack of guidance to exercise. To date, investigating the effect of exercise on sterile inflammation and adapting a lifestyle intervention to SCD - an understudied and minority population - has not been addressed extensively. Therefore, there is a need to develop exercise program for adults with SCD that integrates patient perspectives, is safe, and could modify CV outcomes in SCD. Furthermore, home-based interventions are more accessible, preferred by adults with SCD, and important to widely implementing exercise interventions.18 Our objective is to pilot a home-based exercise intervention tailored for adults with SCD based on patients' preferences. We hypothesize that a moderate-intensity homebased exercise regimen tailored to adults with SCD is feasible and acceptable. The overall long-term objective is to develop a safe exercise intervention to promote sustainable physical activity that could decrease CV risk in SCD.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will include ambulatory adult patients of all SCD genotypes who are in care at UAB's sickle cell center and provide consent to participate in the study.
* Eligible participants include adults with SCD of any genotype older than 18 yrs. of age followed by the UAB sickle cell center.
* Participants must be in steady-state disease defined as not having a vaso-occlusive crisis or SCD-related hospitalization within four weeks of enrollment.

Exclusion Criteria:

* Participants will be excluded if they have severe avascular necrosis of the hip, are pregnant, or have absolute contraindications to exercise according to the American Heart Association (AHA) and American College of Sports Medicine guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility will be measured | One year
  Outcome will be to collect preliminary data on feasibility of the exercise intervention using rates of recruitment and retention

SECONDARY OUTCOMES:
Acceptability will be measured | One year
  Outcome will be to collect preliminary data on acceptability of the exercise intervention using attendance, engagement, and qualitative feedback

OTHER OUTCOMES:
Tolerability will be measured | One year
  Outcome will be to collect preliminary data on tolerability of the exercise intervention using the ability for participants to complete the exercise program without adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Foluso Ogunsile, MD, Principal Investigator — University of Alabama at Birmingham